CLINICAL TRIAL: NCT06807892
Title: CARE-MH: Comparison of Two Cognitive-Motor Rehabilitation Approaches Via Exergames: a Study of Cognitive, Motor and Behavioral Functions in Huntington's Disease Patients
Brief Title: Comparison of Two Cognitive-Motor Rehabilitation Approaches Via Exergames: a Study of Cognitive, Motor and Behavioral Functions in Huntington's Disease Patients
Acronym: CARE-MH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 49RC25_0024
Record Dates: First submitted 2025-01-23; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Huntington's Disease (HD); Exergame

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Synergistic management (Active Comparator)
  Interventions: Other: Synergistic management
- Sequential management (Active Comparator)
  Interventions: Other: Sequential management

INTERVENTIONS:
Other: Synergistic management — In synergistic management, exercises are carried out in a synergistic way: 40 minutes of exercises involving both physical and cognitive stimulation.
  Arms: Synergistic management
Other: Sequential management — In sequential management, exercises are performed sequentially: 20 minutes of physical exercises and 20 minutes of cognitive exercises.
  Arms: Sequential management

SUMMARY:
Huntington's disease (HD) is a rare, hereditary neurodegenerative disorder. It generally manifests itself between the ages of 40 and 50, and results in motor impairment (choreic movements, balance disorders, gait disorders, etc.), cognitive impairment (executive functions, attention, etc.) and behavioral impairment (apathy, depression, irritability, etc.). To date, there is no curative treatment for HD, and drug therapies have little effect on symptomatology, particularly motor symptoms. Physical activity and cognitive stimulation appear to be promising tools in the fight against the progression of various symptoms in certain progressive neurological conditions, including HD. In addition, the use of exergame as an interface is becoming increasingly widespread and offers encouraging prospects in the management of certain neurodegenerative diseases (Parkinson's disease, multiple sclerosis, spinocerebellar ataxia type 3).

The aim of our project is to carry out a preliminary evaluation of the clinical benefit of a management program combining physical activity and cognitive stimulation, compared with a sequential management program.

ELIGIBILITY:
Inclusion Criteria:

* Adults at inclusion
* Huntington's disease diagnosed and confirmed by genetic analysis
* Patient with stage 1-2 HD with a motor UHDRS score ≥ 5 and a CFT between 6 < CFT ≤ 13
* Patient with written informed consent or third-party consent
* Affiliated or beneficiary of a social security scheme

Exclusion Criteria:

* Poor understanding of the French language
* Participation in interventional research modifying management
* History likely to interfere with cognition (established stroke, sequelae of traumatic brain injury, active epilepsy, learning disorders, alcohol dependence syndrome, drug use, psychiatric disorders), severe cognitive deficit (MMSE <16), clinically significant pathological condition which, in the investigator's opinion, could interfere with the subject's safety or the evaluation of study results
* Pregnant or breast-feeding women
* Persons deprived of their liberty by administrative or judicial decision
* Persons under compulsory psychiatric care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-12 (Estimated); Primary Completion 2027-10-17 (Estimated); Study Completion 2027-10-17 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | Sessions are held three times a week for 12 weeks.
  The BBS is a scale comprising 14 tests designed to assess static and dynamic balance. Each test is given a score ranging from 0 (inability to perform the test) to 4 (no difficulty in performing the test), giving a final score out of 56 points (the higher the score, the better the balance skills). The tests included in the BBS are:
  * Sitting
  * Standing without support
  * Standing with feet together
  * Standing with eyes closed
  * From sitting to standing
  * Move from standing to sitting
  * Transfer between two chairs
  * Standing in tandem
  * Stand on one leg
  * Alternating feet on a step or stair while standing
  * Rotate trunk
  * Turn around to look over shoulders
  * Forward movement with arms outstretched
  * Picking up an object from the ground

SECONDARY OUTCOMES:
L'Unified Huntington's Disease Rating Scale - Total Motor Score (UHDRS-TMS) | At the beginning, at the end and 3 months after treatment.
  The UHDRS is the conventional scale for studying the progression of MH symptomatology. It is divided into several subscales grouping together different tests: motor function (vision, dysarthria, dystonia, choreic movements, bradykinesia, walking, etc.), cognitive functions (verbal fluency, Symbol Digit Modalities test, Stroop task, TMT, Digit Memory (WAIS-IV), behavior, functional abilities, independence. For the motor function and behavior subscales, the results are a score, and the higher the score, the greater the motor and behavioral disorders. Conversely, for the cognitive, functional and independence subscales, the higher the score, the stronger the cognitive and functional abilities, and the greater the patient's subjective independence. The UHDRS motor tests are scored from 0 (no impairment) to 4 (severe impairment), giving a total score out of 60 points. The closer the score to 60, the greater the motor impairment.
Six-Minute Walk Test (6MWT) | At the beginning, at the end and 3 months after treatment.
  The 6MWT consists in measuring the distance (in meters) covered in 6 minutes by the participant. It is therefore a recommended tool for measuring walking endurance in MH patients. A straight, flat corridor measuring between 20 and 50 metres is marked out with coloured markers and two cones at either end. The patient is asked to walk as far as possible for 6 minutes, back and forth along the corridor. During the test, the patient can slow down and even stop if necessary, but is obliged to go around the cones at each half-turn. At the end of the 6 minutes, the patient must stop and not move until the distance covered is measured. The longer the total distance covered, the greater the walking endurance.
30 second Chair Stand Test (30CST) | At the beginning, at the end and 3 months after treatment.
  The 30CST consists of standing up and sitting down from a chair as many times as possible for thirty seconds, without physical assistance. The greater the number of repetitions, the greater the muscular strength of the lower limbs.
Mini Mental State Examination (MMSE) | At the beginning, at the end and 3 months after treatment.
  The MMSE enables us to assess global cognitive functioning on a 30-point scale. It comprises 6 subsections: orientation, learning, attention and calculation, recall, language and constructive praxis, scored out of 10, 3, 5, 3, 8 and 1 respectively. The test takes 10 minutes to complete. The higher the score, the better the performance. A score between 22 and 25 suggests mild dementia, between 16 and 20 moderate dementia, between 10 and 15 moderately severe dementia, between 3 and 9 severe dementia and finally very severe dementia below 3. It will be used in this study to check inclusion criteria and assess the patient's overall cognitive abilities.
The working memory subtest of the Wechsler Intelligence Scale for Adults 4th Edition (WAIS-IV, subtest "Number Memory") | At the beginning, at the end and 3 months after treatment.
  The WAIS IV "Digit Memory" sub-test is frequently used in neuropsychological practice to assess auditory attention and auditory working memory. The assessment is carried out in three stages. First, the patient is asked to repeat the digits dictated orally by the evaluator. The exercise starts with 2 digits, and increases after at least one successful attempt out of two. The principle is the same for the next exercise, during which the subject must repeat the sequence of digits in the reverse order to that dictated. For the last exercise, the subject must reconstruct the sequence of numbers in ascending order. Each attempt is marked 0 or 1. The total score is then calculated.
UHDRS cognitive tests - The Stroop test | At the beginning, at the end and 3 months after treatment.
  The Stroop test assesses inhibition. Three boards are presented: the first consists of naming colored rectangles (blue, green or red) and the second of naming words written in letters (blue, green or red). On the third board, the words designating the colors are printed in ink of a different color from that designated. The subject must inhibit reading the word in order to name the ink color.
UHDRS cognitive tests - The Symbol Digit Modalities Test (SDMT) | At the beginning, at the end and 3 months after treatment.
  During the SDMT, which assesses patients' psychomotor speed and working memory, the numbers from 1 to 9 are each associated with a specific symbol on a model. The participant must assign the numbers to the symbols presented line by line. The aim is to correctly associate as many numbers as possible with the different symbols within 90 seconds. The support is written and the model remains in front of the patient for the duration of the test.
UHDRS cognitive tests - Verbal fluency task | At the beginning, at the end and 3 months after treatment.
  The verbal fluency task assessing mental flexibility is composed of two tests: semantic fluency and phonological fluency. In the semantic fluency test, the patient is asked to generate as many words as possible in 1 minute from a category (e.g. fruit, animals, etc.). In the phonological fluency test, the patient is asked to generate a maximum number of words in 1 minute from a letter (e.g. P, R or V).
UHDRS cognitive tests - The Trail Making Test (TMT) | At the beginning, at the end and 3 months after treatment.
  The Trail Making Test is a paper-and-pencil test that assesses spontaneous flexibility. It is offered in two parts. In part A, the subject is asked to connect numbers from 1 to 25 as quickly as possible. For part B, the subject is asked to connect numbers and letters, alternating the number/letter sequence and maintaining ascending numbering and alphabetical order. All stimuli are presented and two examples are performed before each part. Time and errors are recorded.
L'Hospital Anxiety and Depression Scale (HADS) | At the beginning, at the end and 3 months after treatment.
  The Hospital Anxiety and Depression Scale (HADS) is a self-administered questionnaire frequently used to detect anxiety and depressive disorders, common in patients with HD. The self-assessment scale lasts 10 minutes and comprises 14 items (7 for depression and 7 for anxiety) rated from 1 to 3. At the end we then obtain two scores:
  * An anxiety score between 7 and 21. The higher the score, the more severe and disabling the symptoms.
  * A depression score between 7 and 21. The higher the score, the greater and more disabling the symptoms.
Problem Behaviours Assessment for Huntington's Disease (PBA-HD) | At the beginning, at the end and 3 months after treatment.
  The Problem Behaviours Assessment for Huntington's Disease (PBA-HD) is a semi-structured interview questionnaire used to highlight the various behavioural and psychiatric problems that can arise with HD. The original version covers 40 items, but the short version (PBA-s) covers 11 items and evaluates them over the last 4 weeks. Thus, the short version is more commonly used in clinical studies. The 11 items assessed are : Depression; Suicidal ideation; Anxiety; Irritability; Aggressive behavior; Apathy; Perseverative thinking; Obsessive-compulsive disorder; Paranoia; Hallucinations; Disorientation.
  Each item is evaluated with specific questions to produce two types of score:
  * A severity score between 0 and 4. The higher the score, the more severe the symptoms.
  * A frequency score between 0 and 4. The higher the score, the more frequent the symptoms.
SF- 12 self-questionnaire. | At the beginning, at the end and 3 months after treatment.
  The quality of life of patients with HD will be assessed using the SF-12, which is a short version of the SF-36. This is the generic questionnaire most widely used internationally to assess quality of life. It is a 36-question self-administered questionnaire covering eight health domains: the SF-12 consists of 12 questions divided into the same 8 domains as the SF36.
  * Physical functioning
  * Social functioning
  * Limitations due to physical problems
  * Limitations due to emotional problems
  * Mental health
  * Vitality
  * Pain
  * General perception of health For each domain, the scores of the various questions are coded, added together and transformed into a scale ranging from 0 (very poor health) to 100 (very good health).
Acceptance and feasibility | At the beginning, at the end and 3 months after treatment.
  Acceptance and feasibility of the two rehabilitation programs are assessed by the number of sessions completed, the drop-out rate, the rate of correct answers, the rate of early interruption of the session and the duration of the session, as well as by questions on subjective appreciation of the program. Subjective appraisal questions ask patients about the attractiveness of the program (motivation); the clarity, effectiveness and reliability of the exercises (safety); and the hedonic quality (creativity, stimulation) of the program. Patients were asked to answer these questions on a scale from 0 (strongly disagree) to 5 (strongly agree).
  * Do you think the rehabilitation program is attractive (environment, aesthetics)?
  * Do you think the program is effective for your disease?
  * Do you find the information conveyed sufficiently clear (instructions, exercise answers)?
  * Do you feel safe doing the exercises?
  * Are the exercises motivating and stimulating?
Participants' satisfaction | At the beginning, at the end and 3 months after treatment.
  Participants' satisfaction with the program is assessed using a numerical scale: "How would you rate the program and its support overall?" on a scale from 0 (not at all satisfactory) to 5 (completely satisfactory). An open-ended question allows participants to add comments to justify the rating they have received, or to describe how they feel about the program ("Can you justify your rating in a few words, and describe how you feel about the program").

CONTACTS AND LOCATIONS:
Locations (1):
- Angers University hospital, Anngers, France

IPD SHARING:
Plan to Share IPD: No